CLINICAL TRIAL: NCT06651346
Title: Cell-Surface Plectin in the Diagnosis of Cholangiocarcinoma from ERCP-directed Biliary Samples
Status: Not yet recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ross Buerlein, Assistant Professor of Medicine, University of Virginia
Other Study IDs: HSR240084
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cholangiocarcinoma
Keywords: ERCP; Cytology
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cholangiocarcinoma is a malignancy that is most-often diagnosed with ERCP-directed cytology brushings of the biliary tree, but the yield on this cytology has been previously shown to only be 5%-40%. Additionally, the vast majority (approximately 80%) of patients are not diagnosed until they are surgically unresectable (due to late stage at time of diagnosis), at which point there is no chance for cure and their only options are palliative. Therefore, better diagnostic modalities are needed. Plectin is a structural protein located inside of most cells, but it has been shown to be expressed on the cell surface of malignant cells in the pancreaticobiliary tract. The investigators hypothesize that ERCP-guided biliary samples can provide cells and immunohistochemical staining can detect cell surface plectin in patients with cholangiocarcinoma. This would be a novel diagnostic tool which could greatly reduce the time to diagnosis. A previously performed study pilot study at the University of Virginia (unpublished) showed that ERCP-directed biliary biopsies in patients with known cholangiocarcinoma had positive plectin immunohistochemistry, thus showing this is possible. In this current study, patients with a biliary stricture or tumor who are already undergoing ERCP as part of their routine clinical care (i.e. no procedures will be done exclusively for this research study) will undergo an additional biopsy and/or brushing to be assessed for cell-surface plectin expression via immunohistochemistry. The investigators hypothesize that plectin immunohistochemistry will have a higher sensitivity for cholangiocarcinoma than biopsies and/or brushings (cytology) alone.

ELIGIBILITY:
Inclusion Criteria:

* Biliary stricture or mass seen on imaging; already undergoing ERCP as part of their routine clinical care

Exclusion Criteria:

* Age < 18 years old; inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indeterminate biliary strictures or masses who are already undergoing ERCP with biliary tissue sampling in the form of biliary brushings or biopsies
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Positive plectin staining on IHC from ERCP-directed biliary samples | 2 years
  Positive plectin staining on IHC from ERCP-directed biliary samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No